CLINICAL TRIAL: NCT05847309
Title: Optimal Ventilation Time After Endovascular Treatment Under General Anesthesia for Acute Ischemic Stroke. a Prospective, Randomized Comparison Between Early Vs Delayed Extubation
Brief Title: Early Vs Delayed Extubation After Endovascular Treatment for Acute Ischemic Stroke
Acronym: EDESTROKE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Clinico Universitario de Santiago (Other)
Responsible Party: Principal Investigator, Manuel Taboada Muñiz, ASSOCIATE PROFESSOR, Hospital Clinico Universitario de Santiago
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: EDESTROKE
Record Dates: First submitted 2023-04-14; First posted 2023-05-06 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Acute Ischemic Stroke; Endovascular Treatment
Keywords: Stroke; endovascular treatment; Extubation; mechanical ventilation; functional status
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Intervention Model Description: Intervention study, prospective, randomized, parallel and blind for the end point evaluators. (Prospective Randomized, Blinded End-point))
Who Masked: Participant, Investigator
Masking Description: We will compare patients extubated before 6 hours and between 6 to 12 hours after endovascular treatment with general anesthesia for stroke. The patient will not know the hours that he was on mechanical ventilation (masking participant). Investigators evaluating the primary endpoint (mRS at three months) and other secondary endpoints will not know to which group they were randomized. Only the research physicians who treat the patient in the ICU during the first 24 hours know the assigned group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early extubation (Active Comparator): Patients randomized to early extubation, will be extubated < 6 hours after endovascular treatment under general anesthesia.
  Interventions: Other: Early extubation
- Delayed extubation (Experimental): Patients randomized to delayed extubation, will be extubated 6-12 hours after endovascular treatment under general anesthesia.
  Interventions: Other: Delayed extubation

INTERVENTIONS:
Other: Delayed extubation — Patients randomized to delayed extubation, will be extubated 6-12 hours after endovascular treatment under general anesthesia.
  Arms: Delayed extubation
Other: Early extubation — Patients randomized to early extubation, will be extubated < 6 hours after endovascular treatment under general anesthesia.
  Arms: Early extubation

SUMMARY:
Although older studies, most of them retrospective in design, advocated sedation over general anesthesia during endovascular treatment for acute ischemic stroke, a recent meta-analysis and randomized studies have shown that general anesthesia is associated with better functional status at 3 months compared with local anesthesia and sedation. In our center, most procedures are performed under general anesthesia, and once the procedure is complete, the patient is transferred intubated and sedated to the ICU. If the patient is hemodynamically and respiratory stable, the patient will be extubated, and will be discharged to the Neurology hospitalization floor.

Several factors have been described that may influence the evolution and functional status at three months of patients who have suffered a stroke and have received endovascular treatment, such as the time between the onset of symptoms and admission to the ward for performing the procedure, the use of general anesthesia compared to sedation and local anesthesia, adequate control of blood pressure, the size of the cerebral infarct, or a worse neurological examination at the time of the procedure. In turn, several factors have been described that may influence the success of extubation in a patient who has suffered an acute ischemic stroke and who has required orotracheal intubation, such as the absence of dysarthria, the size of the infarct, the location of the infarction, the NIHSS (National Institutes of health Stroke Scale) or neurological status prior to orotracheal intubation. The investigators do not know, however, whether the time of mechanical ventilation can influence the evolution and functional status at three months of patients who have suffered a stroke and have received endovascular treatment under general anesthesia

DETAILED DESCRIPTION:
The authors do not know whether the time of mechanical ventilation can influence the evolution and functional status at three months of patients who have suffered a stroke and have received endovascular treatment under general anesthesia. The purpose of this prospective randomized study is to compare the neurological functional status at 3 months according to the modified Rankin scale (mRS), of patients with stroke who underwent endovascular intervention with satisfactory results and who underwent early extubation (< 6 hours) compared to delayed extubation (6-12 hours).

ELIGIBILITY:
Inclusion Criteria:

* Adult (age ≥ 18 years)
* Acute ischemic stroke due to large intracranial vessel occlusion demonstrated on CT-angiography in the following anterior circulation locations (occlusion of the internal carotid artery and/or middle cerebral artery in segments M1, M2, M3) within 24 hours of symptom onset.
* Patients admitted with a NIHSS neurological status ≥ 6.
* Patients who received endovascular treatment under general anesthesia (intubated in the interventional radiology room) with satisfactory reperfusion (TICI 2b-2c-3).
* Patients admitted in the intensive care unit (ICU) with mechanical ventilation.
* Written informed consent from the patient or proxy (if present) before inclusion or once possible when patient has been included in a context of emergency.

Exclusion Criteria:

* Patients who have not been intubated in the interventional radiology room.
* Pregnancy
* Patients who suffer bronchial aspiration prior to the endovascular procedure or during intubation.
* Patients who underwent the procedure under local anesthesia and sedation.
* Patients with functional neurological status, prior to the ischemic stroke, measured with the modified Rankin scale (mRS) of value: 3-6.
* Patients with vascular involvement of the posterior cerebral circulation, or intracranial haemorrhage associated with stroke.
* Patients who do not sign the informed consent by themselves or their relatives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Modified Ranking Scale (mRS) | 90 days
  Comparison of independent functional outcome as measured by the percentage of patients with a 0 to 2 on the modified Rankin Scale (mRS) at 90 days assessed by study personal blinded to the treatment (early vs delayed extubation)
  The scale of mRS is 0 to 6. The best neurological outcome is the mRS with 0, indicating no any symptom left, and a good neurological outcome is agreed with a mRS 0 to 2. mRS of 6 is the worst, indicating death. mRS will be evaluated by outcome assessor who is blinded to the group

SECONDARY OUTCOMES:
NIHSS (National Institutes of Health Stroke Scale) | Approximately 1-15 days post procedure
  Change in NIHSS score on day 1 and at the time of hospital discharge compared to admission to hospital.
  The NIHSS is composed of 11 items, each of which scores a specific ability between a 0 and 4. For each item, a score of 0 typically indicates normal function in that specific ability, while a higher score is indicative of some level of impairment.The individual scores from each item are summed in order to calculate a patient's total NIHSS score. The maximum possible score is 42, with the minimum score being a 0. NIHSS score of 42 is the worst score (severe stroke), NIHSS score of 0 is "No stroke symptoms".
  0 No stroke symptoms 1-4 Minor stroke 5-15 Moderate stroke 16-20 Moderate to severe stroke 21-42 Severe stroke
Modified Ranking Scale (mRS) | Approximately 3-15 days post procedure
  Comparison of independent functional outcome as measured by the percentage of patients with a 0 to 2 on the modified Rankin Scale (mRS) at the time of hospital discharge assessed by study personal blinded to the treatment (early vs delayed extubation)
  The scale of mRS is 0 to 6. The best neurological outcome is the mRS with 0, indicating no any symptom left, and a good neurological outcome is agreed with a mRS 0 to 2. mRS of 6 is the worst, indicating death. mRS will be evaluated by outcome assessor who is blinded to the group
Hospital length of stay | Approximately 3-15 days post procedure
  Duration in days of hospital stay
Intensive Care Unit length of stay | Approximately 1-15 days post procedure
  Duration in days of ICU stay
Patients extubated in the assigned group | Post procedure within 24 hours
  Percentage of patients who can be extubated in the assigned group
Number of patients with ICU complications | Approximately 1-10 days post procedure
  Complications: Pneumonia, sepsis, bacteraemia, tracheostomy, bronchial aspiration, others
Number of patients with complications associated with mechanical ventilation | Approximately 1-10 days post procedure
  Complications: Pneumonia, pneumothorax, respiratory distress, others
Number of patients with Hospital complications | Approximately 1-15 days post procedure
  Complications: Pneumonia, sepsis, others

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Taboada, Ph.D., Principal Investigator — Clinical University Hospital of Santiago de Compostela; Manuel Rodríguez, M.D., Principal Investigator — Clinical University Hospital of Santiago de Compostela
Locations (1):
- University Clinical Hospital of Santiago de Compostela, Santiago de Compostela, A Coruña, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data types: Deidentified participant data How to access data: Requests must be sent to manutabo@yahoo.es When available: With publication Additional Information Who can access the data: Researchers whose proposed use of the data has been approved Types of analyses: For scientific purpose Mechanisms of data availability: With investigator support
Supporting Information: Study Protocol, SAP, CSR
Time Frame: When available: With publication
Access Criteria: Researchers whose proposed use of the data has been approved Types of analyses: For scientific purpose

REFERENCES:
- [Background] Fandler-Hofler S, Heschl S, Kneihsl M, Arguelles-Delgado P, Niederkorn K, Pichler A, Deutschmann H, Fazekas F, Berghold A, Enzinger C, Gattringer T. Ventilation time and prognosis after stroke thrombectomy: the shorter, the better! Eur J Neurol. 2020 May;27(5):849-855. doi: 10.1111/ene.14178. Epub 2020 Mar 17. PMID 32065457
- [Background] Nikoubashman O, Schurmann K, Probst T, Muller M, Alt JP, Othman AE, Tauber S, Wiesmann M, Reich A. Clinical Impact of Ventilation Duration in Patients with Stroke Undergoing Interventional Treatment under General Anesthesia: The Shorter the Better? AJNR Am J Neuroradiol. 2016 Jun;37(6):1074-9. doi: 10.3174/ajnr.A4680. Epub 2016 Jan 28. PMID 26822729
- [Background] Coplin WM, Pierson DJ, Cooley KD, Newell DW, Rubenfeld GD. Implications of extubation delay in brain-injured patients meeting standard weaning criteria. Am J Respir Crit Care Med. 2000 May;161(5):1530-6. doi: 10.1164/ajrccm.161.5.9905102. PMID 10806150
- [Derived] Taboada M, Estany-Gestal A, Fernandez J, Barreiro L, Williams K, Rodriguez-Yanez M, Otero P, Naveira A, Caruezo V, Veiras S, San Luis E, Dos Santos L, Diaz-Vieito M, Arias-Rivas S, Santamaria-Cadavid M, Rodriguez-Castro E, Vazquez F, Blanco M, Mosquera A, Castineiras JA, Muniategui I, Ferreiroa E, Carinena A, Tubio A, Campana O, Selas S, Aneiros F, Martinez A, Eiras M, Costa J, Prieto JM, Alvarez J. Effect of early vs. delayed extubation on functional outcome among patients with acute ischemic stroke treated with endovascular thrombectomy under general anesthesia: the prospective, randomized controlled EDESTROKE trial study protocol. Trials. 2024 Jun 4;25(1):357. doi: 10.1186/s13063-024-08181-y. PMID 38835061